CLINICAL TRIAL: NCT00725920
Title: Randomized Clinical Trial to Study the Topiramate Efficacy for Posttraumatic Disorder Treatment
Brief Title: Placebo Controled Clinical Trial Using Topiramate To Treat Posttraumatic Stress Disorder (PTSD) Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marcelo Feijo Mello, Associate Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TopirPTSD
Record Dates: First submitted 2008-07-28; First posted 2008-07-31 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD,; posttraumatic; stress; disorder,; randomization,; placebo,; controlled
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Disease | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Experimental): patients receiving the active drug: topiramate
  Interventions: Drug: Topiramate; Drug: placebo control group
- Placebo Control group (Placebo Comparator): patients received pills content placebo, that were identical to the pills content active drug
  Interventions: Drug: placebo control group

INTERVENTIONS:
Drug: Topiramate — patients will receive the active drug. The starting dose was 25 mg/day, with weekly increments of 25 mg/day, according to clinical status. The maximum dose considered was 200 mg/day
  Arms: Topiramate
Drug: placebo control group — initial dose 25 mg day, increments of 25 mg each 2 weeks. Up to 100 mg/day Those with no intolerance and no response dose could be up to 200 mg day
  Other Names: placebo

SUMMARY:
The study is 12-week randomized placebo controlled trial compared to topiramate to treat patients with posttraumatic stress disorder, according to DSM-IV criteria.

Patients will receive topiramate or placebo, the dose will start with 25 mg/day and every week 25mg will be increment according to patients tolerance to side effects.

Patients will be evaluated by blind raters using Clinician-Administered PTSD Scale (CAPS), Beck Depression Inventory (BDI) , Beck Anxiety Inventory (BAI), 36-Item Short Form Health Survey (SF-36), Social Adjustment Scale (SAS).

the outcomes will be improvement on Posttraumatic Stress Disorder (PTSD), Depression, Anxiety, quality of life and social adjustment scale according to scales above.

DETAILED DESCRIPTION:
Seventy-two (72) patients will be randomly allocated, in a stratified manner, according to sex and comorbidity with depression, into two (2) groups: topiramate and routine clinical follow-up, and a group that would receive placebo pills and routine clinical follow-up. The patients will be submitted to evaluations by trained independent researchers, who will apply a structured clinical interview for DSM-IV in order to evaluate the presence of psychiatric disorders (SCID I and SCID-II); the scale of evaluation of the Impact Event Scale-IES; the frequency and intensity of the symptoms of PTSD and of the variations associated with the trauma (PTSD Scale administered by clinical personnel: "Clinician-Administered PTSD Scale" - CAPS); severity of depression: Beck Depression Inventory (BDI) and that of anxiety: Beck Anxiety Inventory (BAI); a scale for the evaluation of social adaptation: Social Adjustment Scale (SAS); a scale for the evaluation of Quality of Life: 36-Item Short Form Health Survey (SF-36) ; a scale for the evaluation of global functioning axis V of DSM-IV (AGF). The patients will receive active treatment for twelve (12) weeks. After this period, the patients who have been using topiramate and who have had an improvement in their clinical condition will continue to receive further treatment for another twelve (12) weeks. Patients will have their medication suspended after twenty four (24) weeks and will be followed-up for a further twenty four (24) weeks. Patients from the placebo group who showed improvement will continue to receive clinical follow-up for a further thirty six (36) weeks. Patients from the placebo group who showed a worsening in their clinical status, evaluated through the CGI, will be excluded from the study and sent for traditional treatment at the PROVE (Violence and Stress Program) clinic. Patients who terminated the active phase of the study who did not obtain a clinical improvement will be sent for traditional treatment at the PROVE clinic. The principal outcomes to be examined will be: Response (a decrease of 50% in the CAPS score starting from the baseline) and remission (lack of diagnostic criteria for PTSD in the CAPS). After the end of the treatment, the collected data will be tabulated and compared using parametric and non-parametric tests. In this study the validation of the CAPS scale for Portuguese will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male and female 18 to 60 yrs old
* PTSD diagnostic according to DSM-IV criteria
* Patients who agree to receive diagnostic after SCID I application by a trained psychiatrist
* Sexually active female patients who agree to use contraceptive
* Patients who agree to sign the IRB approved informed consent

Exclusion Criteria:

* Patients who have schizophrenic disorder, delusional, psychotic depression, schizo-affective, bipolar and dependence to psychoactive substance disorders
* Patients who have clinical disorders not compensated, which require clinical treatment as priority
* Pregnancy
* Previous renal calculosis history
* Being under antidepressant, or other psychotropic medications
* BMI under 20.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-01; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo F Mello, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Mello MF, Yeh MS, Barbosa Neto J, Braga LL, Fiks JP, Mendes DD, Moriyama TS, Valente NL, Costa MC, Mattos P, Bressan RA, Andreoli SB, Mari JJ. A randomized, double-blind, placebo-controlled trial to assess the efficacy of topiramate in the treatment of post-traumatic stress disorder. BMC Psychiatry. 2009 May 29;9:28. doi: 10.1186/1471-244X-9-28. PMID 19480669

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate: patients receiving the active drug: topiramate. Patients will receive topiramate pills, starting at 25 mg/d once daily, at night and increased in 25 mg weekly, as tolerated, until complete or nearly complete efficacy was achieved or until maximum dose allowed was reached (200 mg/d).
- Control Group: patients receiving placebo pills, that were identical to the pills content active drug, starting at 25 mg/d once daily, at night and increased in 25 mg weekly, as tolerated, until complete or nearly complete efficacy was achieved or until maximum dose allowed was reached (200 mg/d).
Period: Overall Study
Arm/Group | Topiramate | Control Group
Started | 17 | 18
Completed | 14 | 12
Not Completed | 3 | 6
Not completed — Lack of Efficacy | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Control Group: patients received pills content placebo, that were identical to the pills content active drug
- Total: Total of all reporting groups
Arm/Group | Topiramate | Control Group | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (13.44) | 36.5 (7.97) | 37.54 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  Brazil | 17 | 18 | 35
Clinician Administered Posttraumatic Scale (CAPS) [Mean (Standard Deviation); unit: scores on a scale]
  Reexperiencing symptoms (CAPS-B) | 23.05 (5.88) | 21.21 (7.15) | 22.84 (3.85)
  Avoidance/numbing symptoms (CAPS-C) | 31.58 (7.13) | 24.78 (11.30) | 28.6 (4.79)
  Hyperarousal symptoms (CAPS-D) | 24.11 (5.69) | 20.14 (8.29) | 22.03 (3.8)
  Total CAPS | 79.64 (12.03) | 64.33 (22) | 72.43 (16.73)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered Posttraumatic Stress Disorder Scale
Description: The Clinician-Administered PTSD Scale (CAPS) [33] : is a structured interview developed to diagnose PTSD and rate its severity. It is comprised of 30-items to assess PTSD-related symptom frequency and severity. Total scores (sum of 3 clusters items) range from 0 to 136, with scores classified as follows: subclinical, from 0 to 19; mild, from 20 to 39; moderate, from 40 to 59; severe, from 60 to 79; extreme, 80 and above.
  CAPS has 3 subscales characterized by the sum of all symptoms for each cluster: CAPS 1 (Revivesce/intrusive recolllections, 5 symptoms, score range: 0-28); CAPS 2 (avoidance, 7 symptoms, score range: 0-36); and CAPS 3 (hyperarousal, 5 symptoms, score range: 0-28).
  CAPS scoring: each symptom scores range from 0 to 4, plus 0-2 scores for frequency, and 0-2 severity.
Time Frame: 12 week
Measure: Mean (Standard Deviation); unit: Total CAPS score
Arm/Group | Topiramate | Control Group
Number analyzed (Participants) | 17 | 18
Total CAPS score | 30.41 (30.90) | 35.78 (33.76)
Statistical Analysis 1: Comparison: Topiramate vs Control Group; Test type: Superiority or Other; p = 0.0076, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Topiramate | Control Group
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 12/17 | 11/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=17) | Control Group (N=18)
somnolence (Nervous system disorders) | 4 (4) | 6 (6)
insomnia (Psychiatric disorders) | 4 (4) | 1 (1)
headache (Nervous system disorders) | 2 (2) | 4 (4)
paresthesia (Nervous system disorders) | 3 (3) | 0 (0)
irritability (Psychiatric disorders) | 2 (2) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
difficulty of concentration (Psychiatric disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes